CLINICAL TRIAL: NCT02668211
Title: Radiostereometric Analysis (RSA) of the PROFEMUR® Preserve Classic Femoral Components
Acronym: TOPAZ
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not feasible - RSA machine not available. RSA images needed for study endpoints
Sponsor: MicroPort Orthopedics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14LJH002
Record Dates: First submitted 2015-11-09; First posted 2016-01-29 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Joint Disease; Osteoarthritis
Keywords: osteoarthritis; radiostereometric analysis; correction of functional deformity; procedures; total hip arthroplasty; musculoskeletal diseases
MeSH Terms: conditions — Joint Diseases; Osteoarthritis; Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PROFEMUR Preserve RSA (Other): Single cohort of subjects prospectively implanted with PROFEMUR® Preserve Classic femoral components
  Interventions: Device: PROFEMUR Preserve Classic Femoral Components

INTERVENTIONS:
Device: PROFEMUR Preserve Classic Femoral Components
  Other Names: Total Hip Arthroplasty System

SUMMARY:
MicroPort Orthopedics (MPO) is conducting this study to investigate the primary stability of its PROFEMUR® Preserve Femoral Components using radiostereometric analysis (RSA). RSA allows precise measurement of micromotion around orthopedic implants and hence, may estimate long-term fixation to bone.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a candidate for primary THA for osteoarthritis
* Subject is able to undergo primary THA procedure
* Subject is a candidate to be implanted with the specified combination of components
* Subject is willing and able to complete required study visits and assessments
* Subject is willing to sign the approved Informed Consent document

Exclusion Criteria:

* Subject has any of the following contraindications at the time of the implantation:
* Overt infection;
* Distant foci of infections (which may cause hematogenous spread to the implant site);
* Rapid disease progression as manifested by joint destruction or bone absorption apparent on roentgenogram;
* Skeletally immature (less than 21 years of age at time of surgery);
* Inadequate neuromuscular status (e.g., prior paralysis, fusion, and/or inadequate abductor strength), poor bone stock, poor skin coverage around the joint which would make the procedure unjustifiable;
* Subjects 76 years of age or older
* Subjects with post-traumatic arthritis in the affected hip
* Subjects with rheumatoid arthritis in the affected hip
* Subjects with hip dysplasia in the affected hip
* Subjects with prior arthroplasty of the affected hip
* Subjects that are morbidly obese (BMI > 35)
* Subjects that are immuno-suppressed
* Subjects with known or tested-positive allergy to metals
* Subjects currently enrolled in another clinical investigation which could affect the endpoints of this protocol
* Subjects unwilling or unable to sign the Informed Consent document
* Subjects with substance abuse issues
* Subjects who are incarcerated or have pending incarceration

Ages: 21 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Assess the stability of the PROFEMUR® Preserve Classic stem with RSA to estimate its long-term performance. | 24 months
  Assessment of the quantity of migration to determine if the total migration of the stem and cup at 2 years post¬operatively are less than 1.2 mm and 2.6mm, and also less than 0.4mm. Assessment of continuous migration to determine if continuous migration, defined as 0.2mm of motion between 1 and 2 years as measured with RSA exists in the stem and cup.
Determine the migration patterns of the PROFEMUR® Preserve Classic stem with RSA | 24 months
  Assessment of migration in each individual plane (x, y, and z), as measured in mm.
Assess if migration pattern is greater than 0.2mm between 1 and 2 years | 24 months
  To determine if the wear rate device is substantially less than the scientifically accepted threshold of 0.1 mm/year for osteolysis. The outcomes will be compared to data from the literature, which states that motion greater than 0.2mm between 1 and 2 years suggests an implant is at risk for early loosening.

SECONDARY OUTCOMES:
Patient functional outcomes (HOOS) | 24 months
  The secondary objective is to determine if there is a significant difference in health status and functional outcomes (using the HOOS questionnaire) before and after total hip arthroplasty (THA) using the PROFEMUR® Preserve Femoral Components.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Maisonneuve Rosemont, Montreal, Quebec, Canada